CLINICAL TRIAL: NCT02036970
Title: A Dose-Ranging Study of the Efficacy and Safety of Bardoxolone Methyl in Patients With Pulmonary Hypertension
Brief Title: Bardoxolone Methyl Evaluation in Patients With Pulmonary Hypertension (PH) - LARIAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 402-C-1302
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension; Interstitial Lung Disease; Idiopathic Interstitial Pneumonia; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Respiratory Bronchiolitis Associated Interstitial Lung Disease; Desquamative Interstitial Pneumonia; Cryptogenic Organizing Pneumonia; Acute Interstitial Pneumonitis; Idiopathic Lymphoid Interstitial Pneumonia; Idiopathic Pleuroparenchymal Fibroelastosis
Keywords: Pulmonary Arterial Hypertension; PAH; Bardoxolone methyl; 6-minute walk distance; CDDO-me; RTA 402; Pulmonary Hypertension; Interstitial Lung Disease; Idiopathic Interstitial Pneumonia; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Respiratory Bronchiolitis Associated ILD; Desquamative Interstitial Pneumonia; Cryptogenic Organizing Pneumonia; Acute Interstitial Pneumonitis; Idiopathic Lymphoid Interstitial Pneumonia; Idiopathic Pleuroparenchymal Fibroelastosis
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Lung Diseases, Interstitial; Idiopathic Interstitial Pneumonias; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Interstitial Pneumonitis, Desquamative, Familial; Cryptogenic Organizing Pneumonia; Hamman-Rich Syndrome | interventions — bardoxolone methyl; ORF 50 transactivator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Part 1 Dose-Ranging Bardoxolone methyl 2.5 mg/Part 2: Open-Label (Experimental): Participants received bardoxolone methyl 2.5 mg once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 continued to receive the same bardoxolone methyl 2.5 mg once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl
- Part 1: Dose-Ranging Bardoxolone methyl 5 mg/Part 2: Open-Label (Experimental): Participants received bardoxolone methyl 5 mg once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 continued to receive the same bardoxolone methyl 5 mg once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl
- Part 1: Dose-Ranging Bardoxolone methyl 10 mg/Part 2: Open-Label (Experimental): Participants received bardoxolone methyl 10 mg once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 continued to receive the same bardoxolone methyl 10 mg once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl
- Part 1: Dose-Ranging Bardoxolone methyl 20 mg/Part 2: Open-Label (Experimental): Participants received bardoxolone methyl 20 mg once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 continued to receive the same bardoxolone methyl 20 mg once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl
- Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone methyl 2.5 mg (Placebo Comparator): Participants received bardoxolone methyl 2.5 mg matching placebo capsules once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 received bardoxolone methyl 2.5 mg once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl; Drug: Placebo
- Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone methyl 5 mg (Placebo Comparator): Participants received bardoxolone methyl 5 mg matching placebo capsules once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 received bardoxolone methyl 5 mg once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl; Drug: Placebo
- Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone methyl 10 mg (Placebo Comparator): Participants received bardoxolone methyl 10 mg matching placebo capsules once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 received bardoxolone methyl 10 mg once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl; Drug: Placebo
- Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone methyl 20 mg (Placebo Comparator): Participants received bardoxolone methyl 20 mg matching placebo capsules once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 received bardoxolone methyl 20 mg once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl; Drug: Placebo
- Part 1: Dose Titration: Bardoxolone methyl 10 mg/Part 2: Bardoxolone methyl 10 mg (Experimental): Participants in Part 1 started with bardoxolone methyl 5 mg once-daily from Day 1 and escalated to bardoxolone methyl 10 mg once-daily starting at Week 4 thru Week 16. Participants who continued to Part 2 continued to receive the same bardoxolone methyl dose once-daily in Part 2 (Week 16 and onwards)
  Interventions: Drug: Bardoxolone methyl
- Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone methyl 10 mg (Placebo Comparator): Participants in Part 1 received Placebo once-daily from Day 1 thru Week 16. Participants who continued to Part 2 initially received bardoxolone methyl 5 mg once-daily from Week 16 thru Week 20 and bardoxolone methyl 10 mg from week 20 onwards
  Interventions: Drug: Bardoxolone methyl; Drug: Placebo

INTERVENTIONS:
Drug: Bardoxolone methyl
  Other Names: RTA 402 capsules
Drug: Placebo
  Arms: Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone methyl 10 mg; Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone methyl 10 mg; Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone methyl 2.5 mg; Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone methyl 20 mg; Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone methyl 5 mg

SUMMARY:
This study assesses the safety and efficacy of bardoxolone methyl relative to placebo in patients with pulmonary hypertension to determine the recommended dose range, evaluate the change from baseline in 6-minute walk distance (6MWD) and determine the effect of Bardoxolone methyl in pulmonary hypertension associated with connective tissue disease, interstitial lung disease, and idiopathic etiologies, including subsets of patients with WHO Group III or WHO Group V PH following 16 weeks of study participation.

DETAILED DESCRIPTION:
The molecular and pharmacological effects of bardoxolone methyl are broad through its induction of Nrf2 and suppression of NF-κB. Bardoxolone methyl may therefore address multiple facets of the pathophysiology of PH because it suppresses activation of proinflammatory mediators, enhances endothelial NO bioavailability, improves metabolic dysfunction, suppresses vascular proliferation, and prevents maladaptive remodeling. Furthermore, while existing therapies primarily target only smooth muscle cells, bardoxolone methyl targets multiple cell types relevant to PH, including endothelial cells, smooth muscle cells, and macrophages.

This is a two-part study.

Part 1: Part 1 of the study will include a dose-ranging phase and a dose-titration phase.

Part 2 (extension period): All patients from Part 1 who complete the 16-week treatment period as planned will be eligible to continue directly into the extension period to evaluate the intermediate and long-term safety and efficacy of bardoxolone methyl.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female patients ≥ 18 to ≤ 75 years of age upon study consent;
2. BMI > 18.5 kg/m²
3. Symptomatic pulmonary hypertension WHO class II and III;
4. WHO Group I, III, or V PH according to the following criteria:

   1. If diagnosed with WHO Group I PAH, then on of the following subtypes:

      * Idiopathic or heritable PAH;
      * PAH associated with connective tissue disease;
      * PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following shunt repair;
      * PAH associated with anorexigen or drug-induced toxicity;
      * PAH associated with human immunodeficiency virus (HIV); or
   2. If WHO Group III PH then primary diagnosis must be one of the following subtypes:

      * Connective tissue disease associated ILD (CTD-ILD);
      * Idiopathic pulmonary fibrosis (IPF);
      * Nonspecific interstitial pneumonia (NSIP); or
   3. If WHO Group V PH then patient must be diagnosed with sarcoidosis;
5. Had a diagnostic right heart catheterization performed and documented within 36 months prior to Day 1 that confirmed a diagnosis of PH
6. If WHO Group I, has been receiving no more than three (3) FDA-approved disease-specific PAH therapies except for intravenous (iv) prostacyclin/prostacyclin analogues. PAH therapy must be at a stable dose for at least 90 days prior to Day 1;
7. Has adequate kidney function defined as an estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73 m2 using the Modification of Diet in Renal Disease (MDRD) 4-variable formula;

Exclusion Criteria:

1. Participation in other interventional clinical studies involving pharmaceutical products being tested or used in a way different from the approved form or when used for an unapproved indication within 30 days prior to Day 1;
2. Initiation of an exercise program for cardio-pulmonary rehabilitation within 3 months (90 days) prior to Day 1 or planned initiation during Part 1 of the study;
3. Stopped receiving any PH chronic therapy within 60 days prior to Day 1;
4. Requirement for receipt of intravenous inotropes within 30 days prior to Day 1;
5. Has uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure (BP) > 160 mm Hg or sitting diastolic blood pressure > 100 mm Hg during Screening after a period of rest;
6. Has systolic BP < 90 mm Hg during Screening after a period of rest;
7. WHO Group III or V patients who at rest require supplemental oxygen at a rate of >4 L/min and have peripheral capillary oxygen saturation levels <92%;
8. Has a history of clinically significant left-sided heart disease and/or clinically significant cardiac disease,including but not limited to any of the following:

   1. Congenital or acquired valvular disease if clinically significant apart from tricuspid valvular insufficiency due to pulmonary hypertension;
   2. Pericardial constriction;
   3. Restrictive or congestive cardiomyopathy;
   4. Left ventricular ejection fraction < 40% per echocardiogram (ECHO) within 60 days of Day 1;
   5. Any current or prior history of symptomatic coronary disease (prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or anginal chest pain);
9. Acutely decompensated heart failure within 30 days prior to Day 1, as per Investigator assessment;
10. History of atrial septostomy within 180 days prior to Day 1;
11. History of obstructive sleep apnea that is untreated;
12. Has a history of portal hypertension or chronic liver disease, including hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication) defined as mild to severe hepatic impairment (Child-Pugh Class A-C);
13. Serum aminotransferase (ALT or AST) levels > the upper limit of normal (ULN) at Screening;
14. For patients with HIV-associated PAH, any of the following:

    1. Concomitant active opportunistic infections within 180 days prior to Screening;
    2. Detectable viral load within 90 days prior to Screening;
    3. Cluster designation (CD+) T-cell count < 200 mm3 within 90 days prior to Screening;
    4. Changes in antiretroviral regimen within 90 days prior to Screening;
    5. Using inhaled pentamidine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-05-31 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (30):
  - Banner University Medical Center, Phoenix Advanced Lung Disease Institute, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Cedars Sinai Medical Center, Beverly Hills, California
  - VA Healthcare System of Greater Los Angeles, Los Angeles, California
  - University of California Davis Medical Center - Division of Pulmonary and Critical Care, Sacramento, California
  - Harbor - UCLA Medical Center, Torrance, California
  - University of Colorado Denver - Division of Pulmonary Sciences, Aurora, Colorado
  - South Denver Cardiology Associates, P.C, Littleton, Colorado
  - Georgetown University Medical Center - Department of Rheumatology, Washington D.C., District of Columbia
  - Cleveland Clinic of Florida, Weston, Florida
  - University of Chicago, Chicago, Illinois
  - Maine Medical Center - Division of Pulmonary and Critical Care Medicine, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai, Beth Israel Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester - University of Rochester Medical Center, Rochester, New York
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University of Cincinnati - Department of Internal Medicine Pulmonary, Critical Care & Sleep Medicine, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - BreatheAmerica El Paso, Inc., El Paso, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - The University of Texas - Health Science Center & Medical School at Houston, Houston, Texas
  - University of Texas Houston - Division of Rheumatology and Clinical Immunogenetics, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Germany (2):
  - University Clinic Carl Gustav Carus, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16). Part 2: Open-label extension period (Week 16 onwards). Part 2 is the extension period and patients were to stay until study drug became available through extended access program [Study 402-C-1602]. Each participant in Part 2 was also in Part 1.
Groups:
- Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label: Participants received bardoxolone methyl 2.5 mg once-daily in Part 1 (Day 1 to Week 16). Participants who continued to Part 2 continued to receive the same bardoxolone methyl 2.5 mg once-daily in Part 2 (Week 16 and onwards)
Period: Part 1: Day 1 Through Week 16
Arm/Group | Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label | Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg | Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg | Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg | Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg
Started | 6 | 12 | 11 | 12 | 2 | 4 | 3 | 4 | 74 | 38
Cohort 1: PAH (BL 6MWD <= 450 Meters) | 6 | 6 | 11 | 6 | 2 | 2 | 3 | 2 | 0 | 0
Cohort 2: PAH (BL 6MWD > 450 Meters) | 0 | 6 | 0 | 6 | 0 | 2 | 0 | 2 | 0 | 0
Cohort 3a: PAH CTD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 8
Cohort 3b: PAH Non-CTD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 9
Cohort 4a: PH CTD-ILD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 8
Cohort 4b: PH CTD-IPF | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
Cohort 4c: PH CTD-IIP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Cohort 4d: PH CTD-Sarcoidosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 1
Completed | 5 | 12 | 7 | 9 | 1 | 3 | 3 | 3 | 66 | 33
Not Completed | 1 | 0 | 4 | 3 | 1 | 1 | 0 | 1 | 8 | 5
Not completed — Adverse Event | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 1 | 3 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 4
Not completed — Progressive Disease | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Week 16 Onwards
Arm/Group | Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label | Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg | Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg | Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg | Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg
Started | 5 | 11 (One patient who completed Part 1 elected not to continue to Part 2.) | 6 (One patient who completed Part 1 elected not to continue to Part 2.) | 9 | 1 | 3 | 3 | 3 | 63 (Three patients who completed Part 1 elected not to continue to Part 2.) | 33
Cohort 1: PAH (BL 6MWD <= 450 Meters) | 5 | 5 | 6 | 5 | 1 | 1 | 3 | 2 | 0 | 0
Cohort 2: PAH (BL 6MWD > 450 Meters) | 0 | 6 | 0 | 4 | 0 | 2 | 0 | 1 | 0 | 0
Cohort 3a: PAH CTD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 8
Cohort 3b: PAH Non-CTD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 7
Cohort 4a: PH CTD-ILD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 7
Cohort 4b: PH CTD-IPF | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Cohort 4c: PH CTD-IIP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Cohort 4d: PH CTD-Sarcoidosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 8
Completed | 5 | 6 | 3 | 7 | 0 | 3 | 2 | 2 | 54 | 28
Not Completed | 0 | 5 | 3 | 2 | 1 | 0 | 1 | 1 | 9 | 5
Not completed — Adverse Event | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 6 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Progressive Disease | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population, which included all randomized patients.
Groups:
- Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 2.5 mg once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 2.5 mg once-daily from Week 16 onwards.
- Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 5 mg once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 5 mg once-daily from Week 16 onwards.
- Part 1: Dose-Ranging Bardoxolone Methly 10 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 10 mg once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 wer eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 10 mg once-daily from Week 16 onwards.
- Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 20 mg once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 20 mg once-daily from Week 16 onwards.
- Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 2.5 mg capsules once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 2.5 mg once-daily from Week 16 and onwards.
- Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 5 mg capsules once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 5 mg once-daily from Week 16 and onwards.
- Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 10 mg capsules once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 10 mg once-daily from Week 16 and onwards.
- Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 20 mg capsules once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 20 mg once-daily from Week 16 and onwards.
- Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg: Part 1: Participants were randomized to receive bardoxolone methyl 10 mg capsules. Participants initially started with bardoxolone methyl 5 mg once-daily from Day 1 and titrated to bardoxolone methyl 10 mg once-daily starting at Week 4 up to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and received the same bardoxolone methyl dose once-daily from Week 16 and onwards.
- Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 10 mg capsules once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 were eligible to continue to the extension Part 2 and initially received bardoxolone methyl 5 mg once-daily from Week 16 thru Week 20 and bardoxolone methyl 10 mg from Week 20 and onwards.
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methly 10 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label | Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg | Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg | Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg | Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg | Total
Number analyzed (Participants) | 6 | 12 | 11 | 12 | 2 | 4 | 3 | 4 | 74 | 38 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed for Part 2 reflects the number of patients who began Part 2 of the study.
  years
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16) | 52.5 (7.15) | 52.8 (14.84) | 50.6 (16.33) | 49.6 (13.06) | 53 (15.56) | 39.5 (11.27) | 54.7 (.58) | 51.3 (8.54) | 56.4 (12.41) | 55.6 (12.7) | 54.3 (12.8)
    Part 2: Open-label extension period (Week 16 and onwards): number analyzed (Participants) | 5 | 11 | 6 | 9 | 1 | 3 | 3 | 3 | 63 | 33 | 137
    Part 2: Open-label extension period (Week 16 and onwards) | 54.6 (5.55) | 53.4 (15.4) | 59.2 (10.26) | 51 (14.76) | 64 (0) | 40 (13.75) | 54.7 (.58) | 47.7 (5.69) | 56.5 (12.23) | 56.7 (12.44) | 55.5 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed for Part 2 reflects the number of patients who began Part 2 of the study.
  Participants
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Female | 4 | 10 | 8 | 11 | 1 | 4 | 2 | 3 | 54 | 27 | 124
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Male | 2 | 2 | 3 | 1 | 1 | 0 | 1 | 1 | 20 | 11 | 42
    Part 2: Open-label extension period (Week 16 and onwards): number analyzed (Participants) | 5 | 11 | 6 | 9 | 1 | 3 | 3 | 3 | 63 | 33 | 137
    Part 2: Open-label extension period (Week 16 and onwards): Female | 4 | 9 | 4 | 9 | 1 | 3 | 2 | 3 | 47 | 24 | 106
    Part 2: Open-label extension period (Week 16 and onwards): Male | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 16 | 9 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed for Part 2 reflects the number of patients who began Part 2 of the study.
  Participants
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Hispanic or Latino | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 12 | 7 | 26
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Not Hispanic or Latino | 4 | 9 | 11 | 11 | 2 | 3 | 3 | 4 | 62 | 31 | 140
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 2: Open-label extension period (Week 16 and onwards): number analyzed (Participants) | 5 | 11 | 6 | 9 | 1 | 3 | 3 | 3 | 63 | 33 | 137
    Part 2: Open-label extension period (Week 16 and onwards): Hispanic or Latino | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 7 | 21
    Part 2: Open-label extension period (Week 16 and onwards): Not Hispanic or Latino | 3 | 9 | 6 | 9 | 1 | 3 | 3 | 3 | 53 | 26 | 116
    Part 2: Open-label extension period (Week 16 and onwards): Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed for Part 2 reflects the number of patients who began Part 2 of the study.
  Participants
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Black or African American | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 17 | 9 | 31
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): White | 6 | 11 | 9 | 12 | 2 | 1 | 3 | 4 | 54 | 28 | 130
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16): Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
    Part 2: Open-label extension period (Week 16 and onwards): number analyzed (Participants) | 5 | 11 | 6 | 9 | 1 | 3 | 3 | 3 | 63 | 33 | 137
    Part 2: Open-label extension period (Week 16 and onwards): American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 2: Open-label extension period (Week 16 and onwards): Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Part 2: Open-label extension period (Week 16 and onwards): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 2: Open-label extension period (Week 16 and onwards): Black or African American | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 14 | 5 | 23
    Part 2: Open-label extension period (Week 16 and onwards): White | 5 | 10 | 5 | 9 | 1 | 0 | 3 | 3 | 47 | 28 | 111
    Part 2: Open-label extension period (Week 16 and onwards): More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 2: Open-label extension period (Week 16 and onwards): Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
6-Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: meters] — Population: Modified Intent-to-treat (mITT) population, which included all randomized patients who received at least 28 doses of study treatment, did not undergo heart or lung transplantation during the treatment period, and performed at least one-post baseline 6MWT assessment. Only Part 1 patients are included since the primary outcome is the change from baseline in 6MWD through Week 16.
  meters | 412 (19.7) | 425.8 (81) | 385.7 (55.45) | 454.5 (93.01) | 358 (96.17) | 418.9 (71.18) | 367 (46.02) | 449.3 (84.64) | 380.8 (96.46) | 395.2 (84.99) | 396.2 (88.32)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Though Week 16 in 6-Minute Walk Distance (6MWD) for Bardoxolone Methyl Compared to Placebo
Description: Overall treatment effect in exercise capacity, as measured by the total distance walked in 6 minutes (6MWD) mean change from baseline though Week 16. A lower 6MWD reflects greater severity thus, a positive change from baseline suggests an improvement.
Time Frame: Baseline through Week 16
Population: mITT population included all randomized patients receiving at least 28 doses of study treatment, did not undergo heart or lung transplantation during the treatment period, and performed at least one-post baseline 6MWD assessment. Only Part 1 patients are included since the primary outcome is the change from baseline in 6MWD through Week 16. Primary outcome assessed for subgroups of participants with PAH from Cohorts 1, 2 and 3 of the study and participants with PH, Cohort 4 of the study.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 10 mg once-daily from Day 1 to Week 16. Part 2: Participants who completed treatment in Part 1 wer eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 10 mg once-daily from Week 16 onwards.
Arm/Group | Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label | Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label | Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg | Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg | Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg | Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg
Number analyzed (Participants) | 6 | 12 | 9 | 10 | 2 | 4 | 3 | 4 | 70 | 38
meters
  Change from Baseline though Week 16 for participants with PAH: number analyzed (Participants) | 6 | 12 | 9 | 10 | 2 | 4 | 3 | 4 | 29 | 17
  Change from Baseline though Week 16 for participants with PAH | 32.5 (29.14) | 24 (30.08) | 3.4 (31.28) | -3.2 (39.53) | 20.3 (13.08) | 24.6 (59.4) | 23.8 (34.54) | -21.8 (4.17) | 13.9 (41.15) | 19.4 (21.06)
  Change from Baseline though Week 16 for participants with PH: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 21
  Change from Baseline though Week 16 for participants with PH |  |  |  |  |  |  |  |  | 7.6 (32.01) | 10.8 (32.01)
Statistical Analysis 1: Comparison: Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label vs Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label vs Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label vs Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label vs Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg vs Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg vs Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg vs Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg vs Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg vs Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg; Overall treatment effect in participants with PAH. Mean overall treatment effect across all visits for change from baseline in 6MWD was estimated and compared with placebo through 16 weeks of treatment using mixed-model repeated measures (MMRM), with treatment group, visit, and the interaction between treatment and visit as fixed factors. A compound symmetry covariance matrix was assumed. Data from Wks 4, 8, 12, and 16 used in the model with the change from baseline at Wk16 as primary endpoint; Test type: Superiority; p = 0.8133, Mixed Models Analysis — The p-value comparison is for the difference in the change in 6WMD from baseline at Week 16 for bardoxolone methyl relative to placebo in participants with pulmonary arterial hypertension (PAH); Mean Difference (Net) = -1.74, 95% CI 2-sided [-16.22 to 12.74] — Mean difference (Net) = Bardoxolone methyl - Placebo
Statistical Analysis 2: Comparison: Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg vs Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg; Overall treatment effect in participants with PH. Mean overall treatment effect across all visits for change from baseline in 6MWD was estimated & compared with placebo through 16 wks of treatment using mixed-model repeated measures (MMRM), with treatment group, visit, and the interaction between treatment & visit as fixed factors. Compound symmetry covariance matrix was assumed. Data from Wks 4, 8, 12, and 16 were used in the model with the change from baseline at Wk 16 as the primary endpoint; Test type: Superiority; p = 0.759, Mixed Models Analysis — The p-value comparison is for the difference in the change in 6WMD from baseline at Week 16 for bardoxolone methyl relative to placebo in participants with pulmonary hypertension (PH); Mean Difference (Net) = -3.17, 95% CI 2-sided [-23.54 to 17.20] — Mean difference (Net) = Bardoxolone methyl - Placebo

ADVERSE EVENTS:
Time Frame: Part 1: 16-week double-blind, randomized, placebo-controlled treatment period (Day 1 to Week 16). Part 2: Open-label extension period (Week 16 onwards). Part 2 is the extension period and patients were to stay until study drug became available through extended access program [Study 402-C-1602].
Groups:
- Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 2.5 mg once-daily from Day 1 to Week 16.
- Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 5 mg once-daily from Day 1 to Week 16.
- Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 10 mg once-daily from Day 1 to Week 16.
- Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label: Part 1: Participants were randomized to receive bardoxolone methyl 20 mg once-daily from Day 1 to Week 16.
- Part 1 Period of Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 2.5 mg capsules once-daily from Day 1 to Week 16.
- Part 1 Period of Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 5 mg capsules once-daily from Day 1 to Week 16.
- Part 1 Period of Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg; Part 1 Period of Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 10 mg capsules once-daily from Day 1 to Week 16.
- Part 1 Period of Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg: Part 1: Participants were randomized to receive bardoxolone methyl matching placebo 20 mg capsules once-daily from Day 1 to Week 16.
- Part 1 Period of Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg: Part 1: Participants were randomized to receive bardoxolone methyl 10 mg capsules. Participants initially started with bardoxolone methyl 5 mg once-daily from Day 1 and titrated to bardoxolone methyl 10 mg once-daily starting at Week 4 up to Week 16.
- Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label: Part 2: Participants who completed treatment receiving bardoxolone methyl 2.5 mg once daily in Part 1 were eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 2.5 mg once-daily from Week 16 onwards.
- Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label: Part 2: Participants who completed treatment receiving bardoxolone methyl 5 mg once daily in Part 1 were eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 5 mg once-daily from Week 16 onwards.
- Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label: Part 2: Participants who completed treatment receiving bardoxolone methyl 10 mg once daily in Part 1 were eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 10 mg once-daily from Week 16 onwards.
- Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label: Part 2: Participants who completed treatment receiving bardoxolone methyl 20 mg once daily in Part 1 were eligible to continue to the extension Part 2 and continued to receive the same bardoxolone methyl 20 mg once-daily from Week 16 onwards.
- Part 2 Period of Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg: Part 2: Participants who completed bardoxolone methyl matching placebo 2.5 mg capsules once-daily treatment in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 2.5 mg once-daily from Week 16 and onwards.
- Part 2 Period of Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg: Part 2: Participants who completed bardoxolone methyl matching placebo 5 mg capsules once-daily treatment in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 5 mg once-daily from Week 16 and onwards.
- Part 2 Period of Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg: Part 2: Participants who completed bardoxolone methyl matching placebo 10 mg capsules once-daily treatment in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 10 mg once-daily from Week 16 and onwards.
- Part 2 Period of Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg: Part 2: Participants who completed bardoxolone methyl matching placebo 20 mg capsules once-daily treatment in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 20 mg once-daily from Week 16 and onwards.
- Part 2 Period of Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg: Part 2: Participants who completed treatment titrated to 10 mg bardoxolone methyl in Part 1 were eligible to continue to the extension Part 2 and received bardoxolone methyl 10 mg once-daily from Week 16 and onwards.
- Part 2 Period of Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg: Part 2: Participants who completed bardoxolone methyl matching placebo 10 mg capsules once-daily treatment in Part 1 were eligible to continue to the extension Part 2 and initially received bardoxolone methyl 5 mg once-daily from Week 16 thru Week 20 and bardoxolone methyl 10 mg from Week 20 and onwards.
Arm/Group | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label | Part 1 Period of Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg | Part 1 Period of Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg | Part 1 Period of Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1 Period of Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg | Part 1 Period of Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 1 Period of Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label | Part 2 Period of Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg | Part 2 Period of Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg | Part 2 Period of Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 2 Period of Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg | Part 2 Period of Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg | Part 2 Period of Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 0/11 | 0/12 | 0/2 | 0/4 | 0/3 | 0/4 | 1/74 | 0/38 | 0/5 | 0/11 | 0/6 | 0/9 | 0/1 | 0/3 | 0/3 | 0/3 | 0/63 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/12 | 0/11 | 2/12 | 0/2 | 0/4 | 0/3 | 1/4 | 7/74 | 2/38 | 2/5 | 5/11 | 3/6 | 6/9 | 0/1 | 1/3 | 2/3 | 1/3 | 9/63 | 9/33
Other Adverse Events (participants affected / at risk) | 5/6 | 11/12 | 10/11 | 12/12 | 2/2 | 4/4 | 3/3 | 4/4 | 64/74 | 33/38 | 5/5 | 11/11 | 6/6 | 8/9 | 1/1 | 2/3 | 3/3 | 3/3 | 50/63 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label (N=6) | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label (N=12) | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label (N=11) | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label (N=12) | Part 1 Period of Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg (N=2) | Part 1 Period of Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg (N=4) | Part 1 Period of Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=3) | Part 1 Period of Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg (N=4) | Part 1 Period of Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=74) | Part 1 Period of Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=38) | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label (N=5) | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label (N=11) | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label (N=6) | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label (N=9) | Part 2 Period of Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg (N=1) | Part 2 Period of Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg (N=3) | Part 2 Period of Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=3) | Part 2 Period of Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg (N=3) | Part 2 Period of Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=63) | Part 2 Period of Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label (N=6) | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label (N=12) | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label (N=11) | Part 1 Period of Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label (N=12) | Part 1 Period of Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg (N=2) | Part 1 Period of Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg (N=4) | Part 1 Period of Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=3) | Part 1 Period of Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg (N=4) | Part 1 Period of Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=74) | Part 1 Period of Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=38) | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 2.5 mg/Part 2: Open-Label (N=5) | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 5 mg/Part 2: Open-Label (N=11) | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 10 mg/Part 2: Open-Label (N=6) | Part 2 Period of Part 1: Dose-Ranging Bardoxolone Methyl 20 mg/Part 2: Open-Label (N=9) | Part 2 Period of Part 1: Dose-Ranging Placebo 2.5 mg/Part 2: Bardoxolone Methyl 2.5 mg (N=1) | Part 2 Period of Part 1: Dose-Ranging Placebo 5 mg/Part 2: Bardoxolone Methyl 5 mg (N=3) | Part 2 Period of Part 1: Dose-Ranging Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=3) | Part 2 Period of Part 1: Dose-Ranging Placebo 20 mg/Part 2: Bardoxolone Methyl 20 mg (N=3) | Part 2 Period of Part 1: Dose Titration: Bardoxolone Methyl 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=63) | Part 2 Period of Part 1: Dose Titration: Placebo 10 mg/Part 2: Bardoxolone Methyl 10 mg (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac discomfort (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scleral disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 3 | 1 | 3 | 0 | 2 | 0 | 1 | 1 | 0 | 4 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 10 | 3 | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 7
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 0 | 1 | 0 | 0 | 10 | 6 | 3 | 4 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 3
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 7 | 4 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 4 | 4
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Implant site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 4 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 5 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Pain (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 7 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 10 | 7 | 2 | 4 | 0 | 1 | 0 | 0 | 1 | 1 | 12 | 9
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 4 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac output increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary arterial pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venous pressure jugular increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vital capacity abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 5 | 1 | 0 | 0 | 0 | 7 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 6
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2 | 1 | 1 | 0 | 0 | 4 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 3 | 0 | 0 | 1 | 0 | 11 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 5 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 4 | 3 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness exertional (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 3 | 5 | 1 | 1 | 1 | 1 | 8 | 7 | 3 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 2 | 3
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 4 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 5 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Digital ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menopause (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT02036970/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT02036970/SAP_001.pdf